CLINICAL TRIAL: NCT01881451
Title: Imaging Tumor Hypoxia With 18F-EF5 PET in Recurrent or Metastatic Clear Cell Ovarian Cancer
Status: Terminated | Type: Observational
Why Stopped: Due to slow accrual and access to the study drug.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Carraressi Foundation OVCARE (Unknown)
Responsible Party: Sponsor
Other Study IDs: H13-00921
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms
Keywords: Tumour hypoxia; Clear Cell Ovarian Cancer; Recurrent; Metastatic
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The collection of archival tumour blocks from the time of prior surgery/biopsy and any newly obtained biopsies (newly obtained biopsies are optional) will be used to construct a tumour tissue microarray (TMA). The TMA will be assessed using multi-parameter staining for LC3A/B (autophagy), EF5 (hypoxia) and cleaved caspase 3 (apoptosis).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 18F-EF5 PET/CT scan — Patients will undergo an investigations 18F-EF5 PET/CT scan.
Procedure: Optional biopsy — Patients who choose to participate, will undergo a tissue biopsy.

SUMMARY:
The purpose of this study is to use 18F-EF5 PET/CT scans to locate areas with low oxygen levels (hypoxia) in patients with recurrent and/or metastatic cancer.

DETAILED DESCRIPTION:
This study involves one visit to the BCCA - Vancouver Centre to undergo one EF5-PET/CT scan. The visit will take about 4 hours to complete and no follow-up visits are required.

* Participants will fill out a short medical questionnaire asking routine information (treatment history, previous surgeries, medications, allergies, etc.) that will take about 5-10 minutes to complete.
* Next they will be weighed and vital signs measured (blood pressure, heart rate and blood oxygen saturation).
* An IV is inserted into a vein in the participant's arm. At the same, a small amount of blood will be taken to measure their blood glucose level.
* The participant will receive an IV dose of 18F-EF5.
* Five minutes after the injection, blood pressure and heart rate will be checked again.
* Participants will then be free to leave the functional imaging department for a period of 180 minutes while the 18F-EF5 circulates throughout their body. Participants are free to eat as normal during this period.
* Participants will undergo the 18F-EF5 PET scan, which will take about 20 minutes. The participant will need to lie still on the scanner bed during the entire scan.
* The 18F-EF5 PET scan will be reviewed by a BC Cancer Agency doctor specialized in PET and the results will be sent to their referring doctor.

Optional Biopsy Procedure:

Participants will have the opportunity of participating in an optional biopsy procedure for the purposes of further studying contemporaneous tumour tissue (contemporaneous with the EF5-PET) for markers of hypoxia, apoptosis, angiogenesis etc. The tissue will also be compared to archival material, and this will allow researchers to study the evolving changes in tumours following treatment.

Patients who consent to undergo a biopsy will be booked to the Diagnostic Imaging Department at the Vancouver Centre. Ultrasound guidance will be used to obtain up to 5 core biopsies from an accessible lesion(s). Up to 2 distinct tumour areas may be sampled. The standard procedure required for a core biopsy will be followed, which will include pre-biopsy lab tests, sterile technique, and when needed, post biopsy observation.

The core biopsies will be formalin fixed and paraffin embedded (FFPE). A BCCA pathologist will review representative slides of each paraffin block to ensure the presence of tumour tissue. The FFPE block will then be sent to the laboratory for immunohistochemistry staining and further interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, advanced metastatic or recurrent clear cell cancer of the ovary
* At least one index lesion measuring 2 cm in diameter
* Must be able to provide written informed consent, and willing to comply with protocol procedures of the study
* Off all active therapy for at least 4 weeks (cytotoxic chemotherapy, radiation, immune therapy, hormone therapy, clinical trials or new agents)

Exclusion Criteria:

* Renal failure (eGFR < 50mls/min)
* Patients with unknown primaries
* Previous history of cancer, except treated non-melanoma skin cancer, non-invasive breast cancer, non-invasive cervical cancer; or curatively treated solid cancer with no evidence of recurrence for more than 5 years.
* Receiving or had received active therapy in the form or chemotherapy or radiation within 4 weeks of the PET scan
* ECOG status ≥ 3
* Unable to tolerate a PET scan which involves an injection of radiopharmaceutical and lying flat and still for 30 minutes.
* Weight more than 204.5 kg (Physical Limitation of Imaging and Radiotherapy Couches) or cannot fit through the PET/CT machine (diameter 70cm).
* Patient is pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants with recurrent or metastatic clear cell ovarian cancer will be approached for study participation at the time of their visit with their treating oncologist (medical oncologist, radiation oncologist or gynecologic oncologist).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Ability of 18F-EF5 to detect areas of tumour hypoxia in clear cell tumours of the ovary | Baseline
  18F-EF5 uptake will be evaluated semi-quantitatively by determining the tumor-to-muscle activity ratio (T/M). Standardized uptake values (SUV) will be calculated for suspicious areas using a region of interest drawn around the target area on the PET images where SUV = (peak activity/mL in region of interest) / (injected activity/g of body weight). A Tumor-to-muscle ratio of >1.5 is considered positive.

SECONDARY OUTCOMES:
Correlate cellular markers of hypoxia and autophagy to the results of the 18F-EF5 PET/CT scans. | Baseline
  Archival tumour tissue will be obtained with consent when possible/available. New biopsies will be obtained as part of the optional consent process, when safe. Archival and new tumour tissue will be assessed using multi-parameter staining for LC3A/B (autophagy), EF5 (hypoxia) and cleaved caspase 3 (apoptosis). Whenever tumour availability is not limited, we will comprehensively assess gene expression involved in hypoxia, angiogenesis, autophagy, apoptosis, and chemotherapy resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tinker, MD, FRCPC, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] GRAY LH, CONGER AD, EBERT M, HORNSEY S, SCOTT OC. The concentration of oxygen dissolved in tissues at the time of irradiation as a factor in radiotherapy. Br J Radiol. 1953 Dec;26(312):638-48. doi: 10.1259/0007-1285-26-312-638. No abstract available. PMID 13106296
- [Background] Fyles AW, Milosevic M, Wong R, Kavanagh MC, Pintilie M, Sun A, Chapman W, Levin W, Manchul L, Keane TJ, Hill RP. Oxygenation predicts radiation response and survival in patients with cervix cancer. Radiother Oncol. 1998 Aug;48(2):149-56. doi: 10.1016/s0167-8140(98)00044-9. PMID 9783886
- [Background] Hockel M, Schlenger K, Knoop C, Vaupel P. Oxygenation of carcinomas of the uterine cervix: evaluation by computerized O2 tension measurements. Cancer Res. 1991 Nov 15;51(22):6098-102. PMID 1933873
- [Background] Evans SM, Hahn SM, Magarelli DP, Zhang PJ, Jenkins WT, Fraker DL, Hsi RA, McKenna WG, Koch CJ. Hypoxia in human intraperitoneal and extremity sarcomas. Int J Radiat Oncol Biol Phys. 2001 Feb 1;49(2):587-96. doi: 10.1016/s0360-3016(00)01494-2. PMID 11173159
- [Background] Nordsmark M, Loncaster J, Aquino-Parsons C, Chou SC, Ladekarl M, Havsteen H, Lindegaard JC, Davidson SE, Varia M, West C, Hunter R, Overgaard J, Raleigh JA. Measurements of hypoxia using pimonidazole and polarographic oxygen-sensitive electrodes in human cervix carcinomas. Radiother Oncol. 2003 Apr;67(1):35-44. doi: 10.1016/s0167-8140(03)00010-0. PMID 12758238
- [Background] Koch CJ, Scheuermann JS, Divgi C, Judy KD, Kachur AV, Freifelder R, Reddin JS, Karp J, Stubbs JB, Hahn SM, Driesbaugh J, Smith D, Prendergast S, Evans SM. Biodistribution and dosimetry of (18)F-EF5 in cancer patients with preliminary comparison of (18)F-EF5 uptake versus EF5 binding in human glioblastoma. Eur J Nucl Med Mol Imaging. 2010 Nov;37(11):2048-59. doi: 10.1007/s00259-010-1517-y. Epub 2010 Jun 29. PMID 20585774
- [Background] Evans SM, Fraker D, Hahn SM, Gleason K, Jenkins WT, Jenkins K, Hwang WT, Zhang P, Mick R, Koch CJ. EF5 binding and clinical outcome in human soft tissue sarcomas. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):922-7. doi: 10.1016/j.ijrobp.2005.05.068. PMID 16458778
- [Background] Evans SM, Judy KD, Dunphy I, Jenkins WT, Hwang WT, Nelson PT, Lustig RA, Jenkins K, Magarelli DP, Hahn SM, Collins RA, Grady MS, Koch CJ. Hypoxia is important in the biology and aggression of human glial brain tumors. Clin Cancer Res. 2004 Dec 15;10(24):8177-84. doi: 10.1158/1078-0432.CCR-04-1081. PMID 15623592
- [Background] Yapp DT, Woo J, Kartono A, Sy J, Oliver T, Skov KA, Koch CJ, Adomat H, Dragowska WH, Fazli L, Ruth T, Adam MJ, Green D, Gleave M. Non-invasive evaluation of tumour hypoxia in the Shionogi tumour model for prostate cancer with 18F-EF5 and positron emission tomography. BJU Int. 2007 May;99(5):1154-60. doi: 10.1111/j.1464-410X.2007.06761.x. Epub 2007 Feb 19. PMID 17309552
- [Background] Komar G, Seppanen M, Eskola O, Lindholm P, Gronroos TJ, Forsback S, Sipila H, Evans SM, Solin O, Minn H. 18F-EF5: a new PET tracer for imaging hypoxia in head and neck cancer. J Nucl Med. 2008 Dec;49(12):1944-51. doi: 10.2967/jnumed.108.053785. Epub 2008 Nov 7. PMID 18997048
- [Background] Mackay HJ, Brady MF, Oza AM, Reuss A, Pujade-Lauraine E, Swart AM, Siddiqui N, Colombo N, Bookman MA, Pfisterer J, du Bois A; Gynecologic Cancer InterGroup. Prognostic relevance of uncommon ovarian histology in women with stage III/IV epithelial ovarian cancer. Int J Gynecol Cancer. 2010 Aug;20(6):945-52. doi: 10.1111/IGC.0b013e3181dd0110. PMID 20683400
- [Background] Spowart JE, Townsend KN, Huwait H, Eshragh S, West NR, Ries JN, Kalloger S, Anglesio M, Gorski SM, Watson PH, Gilks CB, Huntsman DG, Lum JJ. The autophagy protein LC3A correlates with hypoxia and is a prognostic marker of patient survival in clear cell ovarian cancer. J Pathol. 2012 Dec;228(4):437-47. doi: 10.1002/path.4090. PMID 22926683
- [Background] Yamaguchi K, Mandai M, Oura T, Matsumura N, Hamanishi J, Baba T, Matsui S, Murphy SK, Konishi I. Identification of an ovarian clear cell carcinoma gene signature that reflects inherent disease biology and the carcinogenic processes. Oncogene. 2010 Mar 25;29(12):1741-52. doi: 10.1038/onc.2009.470. Epub 2010 Jan 11. PMID 20062075
- [Background] Anglesio MS, George J, Kulbe H, Friedlander M, Rischin D, Lemech C, Power J, Coward J, Cowin PA, House CM, Chakravarty P, Gorringe KL, Campbell IG; Australian Ovarian Cancer Study Group; Okamoto A, Birrer MJ, Huntsman DG, de Fazio A, Kalloger SE, Balkwill F, Gilks CB, Bowtell DD. IL6-STAT3-HIF signaling and therapeutic response to the angiogenesis inhibitor sunitinib in ovarian clear cell cancer. Clin Cancer Res. 2011 Apr 15;17(8):2538-48. doi: 10.1158/1078-0432.CCR-10-3314. Epub 2011 Feb 22. PMID 21343371
- [Background] Stany MP, Vathipadiekal V, Ozbun L, Stone RL, Mok SC, Xue H, Kagami T, Wang Y, McAlpine JN, Bowtell D, Gout PW, Miller DM, Gilks CB, Huntsman DG, Ellard SL, Wang YZ, Vivas-Mejia P, Lopez-Berestein G, Sood AK, Birrer MJ. Identification of novel therapeutic targets in microdissected clear cell ovarian cancers. PLoS One. 2011;6(7):e21121. doi: 10.1371/journal.pone.0021121. Epub 2011 Jul 6. PMID 21754983
- [Background] Cheong H, Lu C, Lindsten T, Thompson CB. Therapeutic targets in cancer cell metabolism and autophagy. Nat Biotechnol. 2012 Jul 10;30(7):671-8. doi: 10.1038/nbt.2285. PMID 22781696
- [Background] Amaravadi RK, Yu D, Lum JJ, Bui T, Christophorou MA, Evan GI, Thomas-Tikhonenko A, Thompson CB. Autophagy inhibition enhances therapy-induced apoptosis in a Myc-induced model of lymphoma. J Clin Invest. 2007 Feb;117(2):326-36. doi: 10.1172/JCI28833. Epub 2007 Jan 18. PMID 17235397
- [Background] Hu YL, DeLay M, Jahangiri A, Molinaro AM, Rose SD, Carbonell WS, Aghi MK. Hypoxia-induced autophagy promotes tumor cell survival and adaptation to antiangiogenic treatment in glioblastoma. Cancer Res. 2012 Apr 1;72(7):1773-83. doi: 10.1158/0008-5472.CAN-11-3831. Epub 2012 Mar 23. PMID 22447568